CLINICAL TRIAL: NCT03990961
Title: Phase II Study of Pembrolizumab for PD-L1 Gene-Altered, Relapsed/Refractory DLBCL
Brief Title: Pembrolizumab for Patients With PD-L1 Diffuse Large B Cell Lymphoma (DLBCL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB19-0076
Record Dates: First submitted 2019-06-17; First posted 2019-06-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-07

CONDITIONS: Diffuse Large B Cell Lymphoma; Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab Treatment (Experimental)
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Subjects will receive pembrolizumab treatment at a dose of 200mg IV every 3 weeks for a duration of 2 years (35 cycles).
  Other Names: Keytruda

SUMMARY:
A non randomized, unblinded, open label phase 2 study to investigate the efficacy of pembrolizumab in patients with relapsed/refractory diffuse large B cell lymphoma (DLBCL) with PD-L1 genetic alterations

ELIGIBILITY:
Inclusion Criteria:

1. Male/female participants who are at least 18 years of age on the day of signing informed consent with a histologically confirmed diagnosis of DLBCL will be enrolled in this study.

   Note: Patients with high-grade B cell lymphomas not otherwised specified and those with MYC and BCL2 translocations (double hit lymphoma) are eligible, as are patients with transformed indolent lymphoma, so long as PD-L1 gene alterations are present.
2. A male participant must agree to use a contraception during the treatment period and for at least 120 days after the last dose of study treatment. Participants must refrain from donating sperm during this period.
3. A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

   1. Not a woman of childbearing potential (WOCBP)
   2. A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 120 days after the last dose of study treatment.

   C.) patient must have negative pregnancy test within 72 hours of beginning treatment if WOCBP
4. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
5. Have measurable disease, defined as at least one lesion that can be accurately measured in at least two dimensions by CT scan. Minimum measurement must be >15 mm in the longest diameter by >10 mm in the short axis. Lesions situated in a previously irradiated area are considered measurable if radiographic progression has been demonstrated in such lesions.
6. Participants must have available archived biopsy material (ideally to be performed shortly before enrollment at the time of most recent relapse) for PD-L1 FISH and correlative studies.
7. There is evidence of a PD-L1 gene alteration within lymphoma cells as assessed by FISH.
8. Participants must have received ≥ 2 lines of prior systemic therapy, ≥ 1 line of prior systemic therapy (if ineligible for or refused autologous stem cell transplantation), or have received 1 line of prior therapy with primary-refractory disease or have relapsed within 12 months from the time of initial diagnosis.

   Note: patients having undergone prior CAR T cell therapy are eligible, as are patients having received a prior allogeneic transplantation, provided they do not meet any of the exclusionary GVHD criteria, and are at least 5 years removed from the date of their transplant.
9. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
10. Have adequate organ function within 10 days prior to the date of treatment allocation. Please see below for Adequate Organ Function Laboratory Values:

    * Hematological

      * Absolute neutrophil count (ANC) less than or equal to 1,000/microliters
      * Platelets less than or equal to 50,000/microliters
      * Hemoglobin less than or equal to 8.0 grams per decilitre
    * Renal

      * Creatinine OR measured or calculated clearance (GFR can also be used in place of creatinine or CrCl) greater than or equal to 1.5XULN OR less than or equal to 30mL/min for participant with creatinine levels less than 1.5 X institutional ULN
    * Hepatic

      * Total bilirubin greater than or equal to 1.5 X ULN or direct bilirubin greater than or equal to ULN for participants with total bilirubin levels less than 1.5 x ULN
      * AST (SGOT) and ALT (SGPT) greater than or equal to 2.5 x ULN (greater than or equal to 5 x ULN for participants with liver metastases)
    * Coagulation

      * International normalized ratio (INR) OR prothrombin time (PT) and Activated partial thromboplastin time (aPTT) greater than or equal to 1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants.

Exclusion Criteria:

1. A WOCBP who has a positive urine pregnancy test within 72 hours prior to treatment allocation . If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
2. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX-40, CD137).
3. Has received chemotherapy, monoclonal antibody therapy, or targeted small molecule therapy within 4 weeks prior to the first dose of study medication. Subjects must have recovered (≤ Grade 1) from adverse events related to a previously administered agent (patients with ≤ Grade 2 neuropathy are eligible). Subjects who have previously received CAR T cell therapy are eligible provided that relapse occurred > 90 days following the date of CAR T cell infusion.

   Note: If a participant received major surgery, he or she must have recovered adequately from complications from the intervention prior to starting study treatment.
4. Has received prior radiotherapy within 1 week of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis.
5. Has a histologic diagnosis of primary mediastinal lymphoma or gray zone lymphoma.
6. Has known active CNS lymphoma and/or lymphomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
7. Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed.
8. Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment.
9. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug. Short courses of corticosteroids will be allowed for palliation of symptoms related to lymphoma, but must be discontinued within 7 days prior to the first dose of study drug.
10. Subjects having received prior allogeneic stem cell transplant, must be at least 5 years removed from the date of their transplant. The also must have no history of severe (grade 3-4) acute GVHD, and/or current > grade 1 acute GHVD. Subjects must not have active chronic GVHD that requires active immune suppression or more than 10 mg of prednisone/day or equivalent.
11. Has a history of a solid organ transplant.
12. Has a known additional malignancy that is progressing or has required active treatment within the past 3 years.

    Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded
13. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
14. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
15. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
16. Has an active infection requiring systemic therapy.
17. Has a known history of Human Immunodeficiency Virus (HIV) infection.
18. Has a known history of Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or known active Hepatitis C virus (defined as detection of HCV RNA) infection.
19. Has a known history of active TB (Bacillus Tuberculosis).
20. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the study, interfere with the subject's participation for the full duration of the study, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
21. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
22. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2023-08-02 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) to pembrolizumab treatment compared to historical controls. | 2 years

SECONDARY OUTCOMES:
Duration of response (DOR) to pembrolizumab treatment | 2 years
Progression-free survival (PFS) | 2 years
Overall survival (OS) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Justin Kline, MD, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago Medicine, Chicago, Illinois, United States